CLINICAL TRIAL: NCT01902121
Title: A Phase 1, Open-label, Randomized, Crossover Clinical Trial in Healthy Normal Volunteers to Evaluate the Bioequivalence of 30 U TI Inhalation Powder Delivered by Gen2 Inhaler Using One 30 U Cartridge Versus a Combination of 10 U and 20 U Cartridges
Brief Title: Compare the Same Dosage of Insulin Using a Combination of Cartridges, 30 Units as 2 Cartridges vs. 1 Cartridge
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MKC-TI-178
Record Dates: First submitted 2013-07-15; First posted 2013-07-18 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TI 30 units (10 unit + 20 unit (Experimental): Technosphere® Insulin 30 units given as 2 cartridges: one 10 unit cartridge + one 20 unit cartridge
  Interventions: Drug: Technosphere® Insulin 10U + 20U
- TI 30 units (30 unit cartridge (Experimental): Technosphere® Insulin 30 units given as one 30 unit cartridge
  Interventions: Drug: Technosphere® Insulin 30U

INTERVENTIONS:
Drug: Technosphere® Insulin 10U + 20U — Inhaled Insulin
  Arms: TI 30 units (10 unit + 20 unit
Drug: Technosphere® Insulin 30U — Inhaled Insulin
  Arms: TI 30 units (30 unit cartridge

SUMMARY:
A Phase 1, open-label, randomized, crossover study in 36 healthy normal volunteers (HNVs) to evaluate the bioequivalence of TI Inhalation Powder delivered using the Gen2 Inhaler and administered as one 30 U cartridge versus a combination of one 10 U cartridge and one 20 U cartridge.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 45 years, considered healthy based on screening physical examination, medical history, clinical chemistry, and urinalysis
* No smoking in the past 6 months (including cigarettes, cigars, and pipes)
* Urine cotinine testing < 100 ng/mL
* Body mass index < 32 kg/m2
* Completion of informed consent form

Exclusion Criteria:

* FBG > 100 mg/dL
* Clinically significant active or chronic illness
* History of asthma, chronic obstructive pulmonary disease (COPD), or any other clinically relevant chronic lung disease
* Respiratory tract infection within 4 weeks before screening and between the screening visit and dosing visit
* Subjects who are experiencing persistent or recurring cough, wheezing, bronchospasm, or dyspnea

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-08; Primary Completion 2013-11 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Area-under-the-serum insulin concentration versus time curve (AUC0-240min | 0, 5, 10, 15, 20, 25, 30, 45, 60, 75, 90, 120, 150, 210 and 240 minutes post-TI dosing

CONTACTS AND LOCATIONS:
Locations (1):
- Neptune City, New Jersey, United States